CLINICAL TRIAL: NCT01745419
Title: Prevalence of Different Haptoglobin Phenotypes in Patients With COPD- Frequent Exacerbators Versus Non Exacerbators
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Michal Steinberg, Dr. Michal Shteinberg, MD, PhD, Carmel Medical Center
Other Study IDs: CMC-12-0121-CTIL
Record Dates: First submitted 2012-12-05; First posted 2012-12-10 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Exacerbation; Haptoglobin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — 3 ml of Serum will be collected from each patient
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD Frequent Exacerbators: COPD patients having experienced at least two episodes of acute exacerbations in the former 12 months. (Acute exacerbations are defined as worsening symptoms requiring treatment with systemic steroids (oral or parenteral) or antibiotics, a visit to the emergency room, and/or admission to a hospital. Events separated by at least 21 days are considered as separate events of exacerbation.)
- COPD non- exacerbators: COPD patients who have not experienced exacerbations in the former 24 months. (Acute exacerbations are defined as worsening symptoms requiring treatment with systemic steroids (oral or parenteral) or antibiotics, a visit to the emergency room, and/or admission to a hospital. Events separated by at least 21 days are considered as separate events of exacerbation.)

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common disease in smokers. COPD has a slowly deteriorating course, punctuated by exacerbations- acute events characterized by increasing shortness of breath and putrid sputum. Exacerbations of COPD may be precipitated by several factors, most commonly infections.

Exacerbation frequency generally increases with declining lung function. However, some patients with COPD consistently experience a higher rate of exacerbations than others despite similar severity of COPD. This has led researchers to postulate the existence of a distinct subgroup of "frequent exacerbators" . Recent work has also brought attention to a subset of patients who experience remarkably few exacerbations despite significantly impaired lung function. Careful characterization of both of these extreme subgroups of COPD may offer additional insights into why certain patients are prone to frequent exacerbations while others remain relatively protected.

Haptoglobin (Hp) is a protein produced predominately by the liver . In humans two types of genes for Hp exist (1 and 2) with possible combinations of these two genes- 1-1, 1-2, or 2-2. The Hp 2 gene is believed to have arisen from the Hp 1 gene in human evolution. Subsequently the prevalence of the Hp 2 allele has spread throughout the world, probably as a result of its ability to provide a selective advantage against infectious disease. The Hp 1-2 combination is a very common one. In most western countries, the prevalence of the Hp genotypes is 16% Hp 1-1, 36% Hp 2-2 and 48% Hp 2-1.

The Hp gene form has been shown to be associated with disease. Specifically, Hp phenotypes have been found to affect propensity to atherosclerosis in Diabetic individuals. There have been several studies suggesting that the Hp 2-2 phenotype is associated with a protection against infectious complications.

In view of the importance of respiratory infections on COPD exacerbations, and of the gained knowledge of Haptoglobin subtypes on propensity to infection, we propose to investigate whether Haptoglobin subtypes are in correlation with the "frequent exacerbator" phenotype of COPD. We postulate that, since people with Hp 1-1 are more prone to infection, the frequency of the Hp 1-1 phenotype will be higher in "frequent exacerbators" of COPD than in "non- exacerbators".

To test our hypothesis we propose to determine Hp phenotype in two groups of COPD patients: one with frequent exacerbations and one with no exacerbations, and compare the relative frequency of the 1-1 phenotype in the two groups.

DETAILED DESCRIPTION:
Laboratory Procedures:

Overview:

3 ml of Serum will be collected and stored at 4 degrees Celsius (up to one week) or minus 20 degrees Celsius until delivery to the laboratory.

Haptoglobin phenotype will be determined at the Department of Anatomy and Cell Biology, the B. Rappaport Faculty of Medicine, 1 Efron st. Haifa, Israel. The method for phenotypin Hp is protein gel electrophoresis.

Serum remaining will be kept frozen in minus 70 degrees Celsius for 5 years in a freezer shelf dedicated for the Pulmonology Institute at the Serology Laboratory in Carmel Medical Center for future analysis of proteins.

Haptoglobin Electrophoresis:

The Haptoglobin protein is separated based on size. Hp 2-2 is the largest therefore was expected to travel the shortest distance in the gel and Hp 1-1 is the smallest and therefore would travel the farthest down the gel. The gel that is used for the electrophoresis was a Polyacrylamide gel. Two concentrations are used in order to provide loading and separating conditions.

The lower gel is a Polyacrilamide gel that contains 10.8 ml 1M Tris pH 8.8, 3.55 ml of Acrylamide 40%, 11.5 ml of dH2O, 225 μl of Ammonium persulfate (APS) 10%, and 18 μl of tetramethylethylenediamine (TEMED). The upper gel is a Polyacrylamide gel that contains 937.5 μl of 1M Tris pH 6.8, 787.5 μl of Acrylamide 40%, 5.7 ml of dH2O, 75 μl of APS 10%, and 7.5 μl of TEMED.

The lower gel is poured in between two glass plates and left for 30 minutes to solidify. Once lower gel is solidified upper gel is poured on top of it, and left for 30 min to solidify. Wells comb placed superiorly to upper gel in order to create wells for sample placement.

The sample for each patient is prepared using 10 μl of the serum, 2 μl of Hemoglobin, and 12 μl of a commercial loading buffer. The sample is then carefully placed in the prepared wells using a pipette. 4 wells are reserved for 3 controls of Hp 2-2, Hp 2-1, and Hp 1-1 followed medially by an empty well.

The western blot analysis is run in a Protean II xi cell by BIO-RAD. The apparatus is assembled and an electrophoresis running buffer is added. The running buffer contains 15.1 g of Tris, 72 g of Glycine, and 1000 ml of DDW. The running buffer was then placed in the upper and lower reservoir of the Protean II. The electrophoresis was run at 240 Volts for 3 hrs.

Once the samples are finished running, the gel is removed from between the glass plates. The gel was then stained using a color staining solution. The Solution was made using 40 mg of 3,3'-5,5' tetramethyl benzidine and 20 ml of methanol. This was left to mix for 15 minutes. Next 2 ml of dimethyl sulfoxide is added and left to mix for 5 min. This was followed by the addition of 40 ml of acetic acid 5% which is made of 2 ml AA and 38 ml of DDW. Next 40 mg of potassium fericyanide dissolved in 4 ml of DDW are added. Finally 600 μl of H2O2 is added to the staining solution and left to mix for 10 min.

Once the staining solution is ready, the gel is placed in a 22 cm by 32 cm tray and the staining solution is poured over the gel. The tray is then placed on a shaker for 25 minutes. Once the Gel is finished being stained it is legible. Nevertheless, the gel is photographed for image enhancement and data storage. The gel is removed from the tray and placed in an Image Analyzer (Imagequant LAS 4000) for imaging, or Canon powershot sx40 hs digital camera.

Data Tabulation:

The data - the Haptoglobin phenotype with corresponding IDs - is gathered and tabulated into a Microsoft excel table.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with COPD according to GOLD guidelines1
2. Age 40-100 years
3. Smoking history of > 10 pack - years
4. Spirometry consistent with airflow obstruction (FEV1/FVC ratio < 70%)
5. Moderate to severe airflow obstruction (FEV1<60%)
6. At least two episodes of acute exacerbations in the former 12 months, or no exacerbations in the former 24 months. (Acute exacerbations are defined as worsening symptoms requiring treatment with systemic steroids (oral or parenteral) or antibiotics, a visit to the emergency room, and/or admission to a hospital. Events separated by at least 21 days are considered as separate events of exacerbation.)

Exclusion Criteria:

Patients with a history of any of the following conditions will be excluded from the study:

1. Active Tuberculosis
2. Pulmonary fibrosis or Asbestosis
3. Organ transplantation
4. Lung volume reduction surgery
5. Previous lung or lobe resection.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of Hp 1-1 phenotype | 1 visit- approximately 2 hours.
  Prevalence as percentage of Hp 1-1 phenotypes in each group of patients

CONTACTS AND LOCATIONS:
Overall Officials: Michal Shteinberg, MD, PhD, Principal Investigator — Pulmonology Institute, Carmel Medical Center
Locations (1):
- Pulmonology Institute, Carmel Medical Center, Haifa, Israel